CLINICAL TRIAL: NCT07237204
Title: A Prospective, Randomized Noninferiority Trial Comparing 15- and 45-minute Pringle Maneuvers During Liver Resection for Oncologic Indications.
Brief Title: 15 vs 45 Minute Pringle Maneuver in Liver Cancer Resection: Randomized Noninferiority Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KB/115/2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Liver Cancer, Adult; Metastases to Liver; Liver Malignant Tumors
Keywords: Pringle manouver; Liver malignancy; Liver resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 minute Pringle manouver with 10 minute reperfusion (Experimental): Hepatic pedicle clamping for 15 minutes, followed by a 10-minute declamping period during liver transection.
  Interventions: Procedure: Pringle manouver
- 45 minute Pringle manouver with 15 minute reperfusion (Experimental): Hepatic pedicle clamping for 45 minutes, followed by a 15-minute declamping period during liver transection.
  Interventions: Procedure: Pringle manouver

INTERVENTIONS:
Procedure: Pringle manouver — The Pringle maneuver involves temporary clamping of the hepatic pedicle during liver resection to reduce blood loss during parenchymal transection.

SUMMARY:
The goal of this clinical trial is to evaluate the safety of two durations of the Pringle maneuver in adults undergoing elective liver resection for malignant tumors. The main questions it aims to answer are:

Is the incidence of post-hepatectomy liver failure different between 15-minute and 45-minute Pringle maneuver durations?

* Do the durations differ in operative time or intraoperative blood loss?
* Researchers will compare patients randomized 1:1 to 15 minutes vs 45 minutes of Pringle clamping to see if outcomes are non-inferior between groups.

Participants will:

* Undergo standard oncologic hepatectomy with the assigned Pringle duration.
* Receive routine perioperative assessments, including laboratory tests and clinical evaluations.
* Attend follow-up visits at approximately 6 months, 1 year, and 3 years after surgery.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria and provide written informed consent will be randomly assigned, using block randomization with a block size of 10, to one of two study groups. In Group 1, Pringle maneuvers lasting 15 minutes with a 10-minute reperfusion interval will be applied during liver resection. In Group 2, Pringle maneuvers lasting 45 minutes with a 15-minute reperfusion interval will be used. In both groups, the Pringle maneuver will be repeated as needed until completion of liver parenchymal transection. If transection is completed earlier, the maneuver will be discontinued before the randomized time. The operating surgeon and anesthesiologist may also decide to start or interrupt the Pringle maneuver outside the predefined time frames if intraoperative conditions require it.

During each Pringle maneuver, the patient's status will be monitored according to standard practice for liver resection, including blood pressure measurement, urine output, and arterial blood gas analysis. The number and duration of Pringle maneuvers, arterial blood pressure values, the type and doses of vasopressors used, serum lactate levels, the duration of parenchymal transection, total operative time, intraoperative blood loss, and hourly urine output will be recorded in perioperative case report forms.

In the postoperative period, laboratory tests will be performed on postoperative days 0, 1, 3, and 5. The occurrence of postoperative complications up to the time of hospital discharge will be documented in the patient's electronic medical record. Outcomes will be assessed by in-person outpatient visits or telemedicine consultations at approximately 6 months, 1 year, and 3 years after surgery.

The sample size was calculated using the Wald method. Based on an analysis of archival data from the Department of Transplantation and Liver Surgery, the incidence of post-hepatectomy liver failure according to the ISGLS definition is approximately 4%. Assuming 80% power, a one-sided significance level of 0.05, and a noninferiority margin of 5%, 300 participants will be enrolled in each arm.

Collected study data will be analyzed with particular attention to the duration of the Pringle maneuver, the extent and technical complexity of the resection, the primary diagnosis, and the presence of coexisting liver disease, in order to determine their influence on the study endpoints.

An interim analysis is planned after recruitment of 50% of the target sample size. If the interim analysis demonstrates a negative effect of the intervention on postoperative complications, further enrollment will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a primary or secondary malignant liver tumor.
* Age > 18 years.
* Patient deemed eligible for liver resection.
* WHO performance status ≤ 2.
* Ability to provide written informed consent.

Exclusion Criteria:

* Liver cirrhosis.
* Liver dysfunction classified as Child-Pugh class B or C.
* Repeat hepatectomy.
* Prior ablation or chemoembolization of hepatic lesions.
* Prior portal vein branch embolization.
* Planned or performed ALPPS procedure.
* Concomitant resection of any organ other than the gallbladder during the same operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Posthepatectomy liver failure | On or after postoperative day 5
  Posthepatectomy liver failure defined by the International Study Group of Liver Surgery as a postoperative deterioration of the liver's synthetic, excretory, and detoxifying functions, characterized by an increased INR and concomitant hyperbilirubinemia (per local lab normals) on or after postoperative day 5.

SECONDARY OUTCOMES:
Intraoperative blood loss | At the completion of the surgery
  Intraoperative blood loss is the volume of blood lost during surgery, calculated as the total volume in the suction canister(s) minus the volume of irrigation fluid administered during the procedure.
Parenchymal transection time | At the completion of the surgery
  Time elapsed from the start of liver parenchymal transection to completion of parenchymal transection.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Kruk, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD). The design of this study does not require public IPD sharing for the reliability of the published results. De-identified IPD may be provided to journal peer reviewers under confidentiality during manuscript review.

REFERENCES:
- [Background] Wang HP, Hou TY, Li WF, Yong CC. Inflow control can be safely used in laparoscopic subsegmentectomy of the liver: a single-center 10-year experience. BMC Surg. 2023 Dec 6;23(1):366. doi: 10.1186/s12893-023-02282-2. PMID 38057769
- [Background] van den Broek MA, Bloemen JG, Dello SA, van de Poll MC, Olde Damink SW, Dejong CH. Randomized controlled trial analyzing the effect of 15 or 30 min intermittent Pringle maneuver on hepatocellular damage during liver surgery. J Hepatol. 2011 Aug;55(2):337-45. doi: 10.1016/j.jhep.2010.11.024. Epub 2010 Dec 13. PMID 21147188
- [Background] Doi S, Yasuda S, Hokuto D, Kamitani N, Matsuo Y, Sakata T, Nishiwada S, Nagai M, Nakamura K, Terai T, Kohara Y, Sho M. Impact of the Prolonged Intermittent Pringle Maneuver on Post-Hepatectomy Liver Failure: Comparison of Open and Laparoscopic Approaches. World J Surg. 2023 Dec;47(12):3328-3337. doi: 10.1007/s00268-023-07201-3. Epub 2023 Oct 3. PMID 37787778
- [Background] Liu J, Wang W, Shi C, Li C, Xue F, Hu L, Wang Y, Ge R. The difference in prolonged continuous and intermittent Pringle maneuver during complex hepatectomy for hepatocellular carcinoma patients with chronic liver disease: A retrospective cohort study. Cancer Med. 2021 Dec;10(23):8507-8517. doi: 10.1002/cam4.4361. Epub 2021 Oct 18. PMID 34658153
- [Background] Fagenson AM, Gleeson EM, Nabi F, Lau KN, Pitt HA. When does a Pringle Maneuver cause harm? HPB (Oxford). 2021 Apr;23(4):587-594. doi: 10.1016/j.hpb.2020.07.014. Epub 2020 Sep 12. PMID 32933844
- [Background] Huang Y, Liao A, Pu X, Yang J, Lv T, Yan L, Yang J, Wu H, Jiang L. A randomized controlled trial of effect of 15- or 25-minute intermittent Pringle maneuver on hepatectomy for hepatocellular carcinoma. Surgery. 2022 Jun;171(6):1596-1604. doi: 10.1016/j.surg.2021.11.012. Epub 2021 Dec 13. PMID 34916072